CLINICAL TRIAL: NCT06723769
Title: Efficacy and Safety of Low-frequency Repetitive Transcranial Magnetic Stimulation in Post-stroke Depression: a Randomized Controlled fNIRS Study
Brief Title: Efficacy of Repeated Transcranial Magnetic Stimulation Based on Near-infrared Imaging in Patients With Post-stroke Depression
Acronym: PSD fNIRS rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dingqun Bai (Other)
Responsible Party: Sponsor-Investigator, Dingqun Bai, Director of rehabilitation Medicine, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20241204
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Post-stroke Depression
Keywords: fNIRS; LF-rTMS; DLPFC
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): conventional treatment
  Interventions: Other: conventional treatment
- rTMS group (Experimental): The rTMS group was treated with LF-rTMS based on the conventional treatment.
  Interventions: Device: rTMS treatment

INTERVENTIONS:
Device: rTMS treatment — Repetitive transcranial magnetic stimulation (rTMS) is a new physiotherapy technique for the treatment of PSD Compared to other strategies, it has the advantages of simple operation, non-invasive, painless, and safe. Studies have comprehensively shown that rTMS can effectively improve depressive symptoms in PSD patients
  Arms: rTMS group
Other: conventional treatment — general treatment of stabilizing vital signs (such as antidepressants, stabilizing blood pressure, stabilizing blood sugar, etc. ) and conventional rehabilitation treatment (hemiplegic limb comprehensive training, swallowing speech training, cognitive perception training, etc. ).
  Arms: Control group

SUMMARY:
This is a randomized controlled trial to evaluate the efficacy and safety of Low-frequency repetitive transcranial magnetic stimulation (LF-rTMS) in post-stroke depression (PSD), explore mechanism of rTMS with Functional near-infrared spectroscopy (fNIRS).

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of low-frequency repetitive transcranial magnetic stimulation (LF-rTMS) for the right dorsolateral prefrontal cortex (DLPFC) in patients with post-stroke depression (PSD), and explore the possible neural mechanism of rTMS with Functional near-infrared spectroscopy (fNIRS).

Patients were randomly assigned to the rTMS and control groups. the treatment effect was assessed by the Hamilton Depression Scale (HAMD), Hamilton Anxiety Scale (HAMA), National Institutes of Health Stroke Scale (NIHSS), and Barthel Index (BI). Meanwhile, fNIRS was used to detect the changes of blood oxygen concentration in the frontal cortex.

After treatment, the score of the HAMD scale in the rTMS group decreased more significantly than in the control group (P<0.05). The value of CH17 oxyhemoglobin (HBO) and the value of CH6 deoxyhemoglobin (HBR) were decreased after rTMS. The HbR of CH6 and CH8 decreased significantly, the HbR of CH12 and CH15 increased significantly (P<0.05). The HAMA, NIHSS and Barthel scores improved more significantly in the rTMS group.

ELIGIBILITY:
Inclusion Criteria:

* 1) Hospitalized patients over 18 years of age; (2) Meet the stroke diagnostic criteria of the Fourth National Conference on Cerebrovascular Diseases and have been confirmed as ischemic or hemorrhagic stroke by head CT and MRI; (3) Symptoms of PSD such as low mood, loss of interest in daily life, insomnia, or poor appetite persist for more than 1 week and meet the inclusion criteria of the DSM-5; (4) Hamilton Depression Scale score-17 (HAMD) > 7; (5) Stable vital signs, willing to accept the treatment method of this study, and sign the informed consent for treatment.

Exclusion Criteria:

* (1) Patients with a history of mental disorders and depression before stroke onset; (2) Patients with consciousness disorder, severe aphasia or comprehension and expression disorder after stroke; (3) Patients with serious cognitive impairment can not cooperate with the psychological evaluator; (4) Patients with metal implants in the skull; (5) People with cardiac pacemakers; (6) Previous head trauma, alcoholism, or family history of epilepsy and another risk of seizures; (7) psychotic symptoms such as agitation, speech and behavior disorder; (8) refuse to sign the informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale (HAMD-17) | pre and post 4 weeks treatment
  evaluate the degree of depression
Functional near-infrared spectroscopy (fNIRS assessment) | pre and post 4 weeks treatment
  measure brain function to determine the effect of rTMS on cerebral blood flow change

SECONDARY OUTCOMES:
Hamilton Anxiety Scale(HAMA) | pre and post 4 weeks treatment
  evaluate the degree of anxiety
National Institutes of Health Stroke Scale(NIHSS) | pre and post 4 weeks treatment
  evaluate the degree of neurological impairment
Barthel Index(BI) | pre and post 4 weeks treatment
  evaluate the degree of daily living ability

CONTACTS AND LOCATIONS:
Overall Officials: Dingqun Bai, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- Department of Rehabilitation Medicine, the First Affiliated Hospital of Chongqing Medical University, Chongqing,, Chongqing, Chongqing 400010, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided